CLINICAL TRIAL: NCT02059369
Title: Ablation of Complex Fractionated Electrograms With or Without Additional Linear Lesions for Persistent Atrial Fibrillation
Acronym: ADLINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-013
Record Dates: First submitted 2013-05-23; First posted 2014-02-11 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation; Recurrence
Keywords: Atrial fibrillation; Recurrence; CFAE; linear ablation
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CFAE ablation (Active Comparator): Intervention: Complex fractionated atrial electrograms (CFAE) Ablation
  Interventions: Procedure: PVI+CFAE+DCC
- CFAE + Lines (Active Comparator): CFAE Ablation followed by linear lesions (anterior and Roof line)
  Interventions: Procedure: PVI, CFAE, anterior and roof line, DCC

INTERVENTIONS:
Procedure: PVI+CFAE+DCC — pulmonary vein Isolation (PVI), CFAE for substrate modification and direct current cardioversion (DCC) if AF persists
  Arms: CFAE ablation
Procedure: PVI, CFAE, anterior and roof line, DCC — PVI, CFAE ablation. If AF persists linear lesions (anterior and roof line), cardioversion if AF persists
  Arms: CFAE + Lines

SUMMARY:
While there is a consensus to perform pulmonary vein isolation (PVI) as a cornerstone for paroxysmal and persistent atrial fibrillation (AF), different additional ablation approaches are used for substrate modification: linear lesions, ablation of complex fractionated atrial electrograms (CFAE) or a combination of both. The aim of this study is to determine whether there is a difference in terms of freedom from arrhythmia recurrence between PVI with CFAE ablation in combination or not with linear lesions in patients with persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic persistent AF
* After PVI +CFAE ablation, no termination into sinusrhythm or atrial tachycardia

Exclusion Criteria:

* Left atrial thrombus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Freedom from atrial arrhythmia | 12 months
  Documented freedom from atrial arrhythmia (AF or AT) recurrence

SECONDARY OUTCOMES:
Procedural and safety data | 12 months
  Duration of procedure, ablation time, fluoroscopy time and complications
Number and result of reablation procedure | 12 months
  Number of redo procedures, results and type of recurrent arrhythmia

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum München, Munich, Germany